CLINICAL TRIAL: NCT01916096
Title: Lancet Blood Volume Comparison Study
Status: Completed | Type: Observational
Sponsor: Facet Technologies (Other)
Responsible Party: Sponsor
Other Study IDs: FT-837-068-BV
Record Dates: First submitted 2013-08-01; First posted 2013-08-05 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Delica 28g Depth 3 vs Delica 30g Depth 3: 30 subjects with diabetes
  Interventions: Device: Delica Device
- Delica 28g Depth 5 vs Delica 30g Depth 5: 30 subjects with diabetes
  Interventions: Device: Delica Device
- Delica 28g Depth 7 vs Delica 30g Depth 7: 30 subjects with diabetes
  Interventions: Device: Delica Device
- Delica 28g Depth 3 vs Delica 33g Depth 3: 30 subjects with diabetes
  Interventions: Device: Delica Device
- Delica 28g Depth 5 vs Delica 33g Depth 5: 30 subjects with diabetes
  Interventions: Device: Delica Device
- Delica 28g Depth 7 vs Delica 33g Depth 7: 30 subjects with diabetes
  Interventions: Device: Delica Device

INTERVENTIONS:
Device: Delica Device

SUMMARY:
The primary objective of the study examines the success rate of various OneTouch Delica lancet sizes across depth settings of the OneTouch Delica lancing device. The sample size is based on 30 subjects per lancet size for a given depth setting. Each subject is lanced 4 times with two lancet sizes at a single depth setting. There will be 120 paired lancing events for each lancet size within the group.

Null hypothesis (H0): there is a 90% success rate of attaining a minimum blood volume of 1.0μL for the 28g lancet across all depth settings.

Alternate hypothesis (H1): the success rate of attaining a minimum blood volume of 1.0μL for the 28g lancet across all depth settings is less than 90%.

ELIGIBILITY:
Inclusion Criteria:

* Must have been diagnosed with type 1 or type 2 diabetes for at least 1 year
* Must be doing Blood Glucose Monitoring, at least twice daily for at least 6 months
* Subjects must be between 18 and 85 years of age.
* Subjects must be able to perform all tasks required in this protocol.
* Subjects must be willing to complete all study procedures.
* Subjects must be able to speak, read and understand English and understand the Informed Consent document.

Exclusion Criteria:

* Subjects with neuropathy or any other nerve damage in the hand or fingers
* Subjects who are taking prescription anti-coagulants or more than one full aspirin per day during the past week or have clotting problems that may prolong bleeding (persons taking Plavix or a daily low dose aspirin will not be excluded but this will be recorded).
* Subjects taking prescription medications for neuropathy.
* Subjects with hemophilia or any other bleeding disorder.
* Subjects with infection with a blood borne pathogen (e.g., HIV, hepatitis).
* Subjects having a condition such as a cognitive disorder, which in the opinion of the Investigator would put the person at risk or seriously compromise the integrity of the study (PI will sign case report form if subject is excluded).
* Subjects working for Facet, LifeScan Inc., or a competitive company.
* Subjects with missing digits.
* Subjects who are pregnant or nursing.
* Subjects on chemotherapy.
* Subjects with poor circulation to the hands as judged by a refill time of more than 5 seconds

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with diabetes from the surrounding communitu
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2012-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Blood Volume Measurements | 24 hours
  Lancing events were performed on subjects fingers. After each lancing event blood volume was measure with a scale.

CONTACTS AND LOCATIONS:
Overall Officials: Barry Ginsberg, MD, Study Chair — Facet Technologies
Locations (1):
- Facet Technologies, Kennesaw, Georgia, United States